CLINICAL TRIAL: NCT04509570
Title: A Prospective & Retrospective Study on the Presence of Ectopic Lymphoid-like Structures and Intralesional Steroid Injection for the Chronic Skin Lesion of Autoimmune Bullous Disease Patients
Brief Title: A Prospective & Retrospective Study on Ectopic Lymphoid-like Structures in Chronic Skins of Autoimmune Bullous Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Jong Hoon Kim, MD, PhD, Associate Professor, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-2018-0302
Record Dates: First submitted 2020-07-28; First posted 2020-08-12 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Autoimmune Bullous Disease
Keywords: ELS
MeSH Terms: interventions — Biopsy; Steroids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment: ILI(Intralesional injection) (Other): 5~20mg/ml, intralesional injection every 1 month. Number of cycles: until the lesions are clinically cleared
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — 5~20mg/ml, intralesional injection every 1 month. Number of cycles: until the lesions are clinically cleared
  Other Names: Steroid injection

SUMMARY:
The purpose of this study is to identify the presence or absence of ectopic lymph node-like structures in skin lesions of patients with autoimmune bullous disease and the subtypes of the cells deposited there. In addition, this study clarifies the therapeutic effect of intralesional steroid injection in patients with pemphigus harboring ectopic lymph node-like structure.

ELIGIBILITY:
Inclusion Criteria:

<Presence of Ectopic Lymphoid-like Structures in the Skin lesion of Autoimmune Bullous Disease Patients>

Prospective study Inclusion Criteria:

1. Adults over 19
2. Patietns who voluntarily signed the consent form
3. Patients who are diagnosed with autoimmune bullous disease through clinical, histological and serological tests

Retrospective study Inclusion Criteria:

1. Samples in human-derived banks from March 2013 to October 2018
2. Patients who are diagnosed with autoimmune bullous disease through clinical, histological and serological tests
3. Adults over 19 <Treatment of Ectopic Lymphoid-like Structures in the Skin lesion of Autoimmune Bullous Disease Patients>

Prospective study Inclusion Criteria:

1. Adults over 19
2. Patients who voluntarily signed the consent form
3. Patients who have skin lesions harboring ectopic lymph node-like structure in a prospective or retrospective manner
4. Patients who have chronic lesions sustained for more than 4 months during the treatment of systemic corticosteroids

Retrospective study Inclusion Criteria:

1. Patients who have skin lesions harboring ectopic lymph node-like structure in a retrospective manner
2. Paitents who have been treated for intralesional steroid injection
3. Patients who have data of photography to compare the clinical effects before and after intralesional corticosteroid treatment.

Exclusion Criteria:

1. Patients who do not meet the criteria for autoimmune bullous disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Clinical outcome: size of lesions | through study completion, an average of 1 year
  The area of the lesions will be measured using the Image J program

SECONDARY OUTCOMES:
The presence or absence of ectopic-lymph node-like structure by histologic evaluation | through study completion, an average of 1 year
  The presence of absence of ectopic-lymph node-like structure will be evaluated by histologic evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Han D, Lee AY, Kim T, Choi JY, Cho MY, Song A, Kim C, Shim JH, Kim HJ, Kim H, D'Angio HB, Preska R, Mayer AT, Kim M, Choi EJ, Kim TG, Shin EC, Park K, Kim DY, Kim SC, Kim JH. Microenvironmental network of clonal CXCL13+CD4+ T cells and Tregs in pemphigus chronic blisters. J Clin Invest. 2023 Dec 1;133(23):e166357. doi: 10.1172/JCI166357. PMID 37815865